CLINICAL TRIAL: NCT06858579
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study To Evaluate The Efficacy And Safety Of DNTH103 In Adults With Chronic Inflammatory Demyelinating Polyneuropathy (CAPTIVATE)
Brief Title: A Study to Evaluate the Efficacy and Safety of DNTH103 in Adults With Chronic Inflammatory Demyelinating Polyneuropathy (CAPTIVATE)
Acronym: CAPTIVATE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dianthus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DNTH103-CIDP-301; 2024-517529-26 (Other: EU CT Number)
Record Dates: First submitted 2025-02-18; First posted 2025-03-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- DNTH103 (Part A) (Experimental): DNTH103 intravenous (IV) loading dose on Day 1.
  DNTH103 subcutaneous (SC) once every 2 weeks for up to 13 weeks.
  Interventions: Drug: DNTH103
- DNTH103 Low Dose (Part B) (Experimental): DNTH103 SC once every 2 weeks for up to 52 weeks.
  Interventions: Drug: DNTH103
- DNTH103 High Dose (Part B) (Experimental): DNTH103 SC once every 2 weeks for up to 52 weeks.
  Interventions: Drug: DNTH103
- Placebo (Part B) (Placebo Comparator): Placebo SC once every 2 weeks for up to 52 weeks.
  Interventions: Drug: Placebo
- DNTH103 (Optional OLE) (Experimental): DNTH103 SC once every 2 weeks for up to 104 weeks.
  Interventions: Drug: DNTH103

INTERVENTIONS:
Drug: DNTH103 — IV Infusion
  Other Names: Claseprubart
  Arms: DNTH103 (Part A)
Drug: DNTH103 — SC injection
  Other Names: Claseprubart
  Arms: DNTH103 (Optional OLE); DNTH103 (Part A); DNTH103 High Dose (Part B); DNTH103 Low Dose (Part B)
Drug: Placebo — SC injection
  Arms: Placebo (Part B)

SUMMARY:
The purpose of this Phase 3 study is to demonstrate the efficacy of DNTH103 as compared to placebo in participants with chronic inflammatory demyelinating polyneuropathy (CIDP).

DETAILED DESCRIPTION:
The study includes the following periods:

* Part A: An open-label period (up to 13 weeks)
* Part B: A randomized, placebo-controlled, double-blind treatment period (up to 52 weeks) for participants who respond to DNTH103 in Part A
* Optional open-label extension (OLE) for eligible participants (up to 104 weeks)
* Safety follow-up (40 weeks)

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out.
2. Weight range between 40 kilograms (kg) and 120 kg.
3. Confirmed diagnosis of CIDP or possible CIDP. Participants must have either typical CIDP or one of the following variants: motor or multifocal CIDP. Diagnosis must be confirmed by the Independent CIDP Review Panel.
4. CIDP Disease Activity Status (CDAS) score ≥ 3 at screening.
5. Must be neurologically stable.
6. Must have an INCAT score between 2 and 9 inclusive.
7. Must fulfill one of the following treatment conditions for CIDP:

   1. Currently treated with and responded to immunoglobulin (Ig) (intravenous immunoglobulin [IVIg] or subcutaneous immunoglobulin [SCIg]) alone or Ig (IVIg or SCIg) plus oral corticosteroids, or previously treated with and responded to, but are no longer being treated with (eg, lost access to), a maintenance regimen of Ig (IVIg or SCIg) alone or Ig (IVIg or SCIg) plus oral corticosteroids.
   2. Currently treated with and responded to oral corticosteroids alone or oral corticosteroids in combination with azathioprine or mycophenolate mofetil.
   3. Refractory participants who have had treatment failure (worsening) or an inadequate response to Ig and/or oral corticosteroids (defined as no clinically meaningful improvement after a period of a minimum of 12 weeks, which may include both active treatment and observation to assess response), or who at any time were unable to tolerate these treatments, experienced adverse effects, or have documented contraindications.
   4. Treatment naïve with no history of prior treatment for CIDP.
8. Documented vaccinations against encapsulated bacteria in accordance with local requirements and vaccine availability.
9. Female participants must be of nonchildbearing potential or if of childbearing potential, must agree not to donate ova, not to attempt to become pregnant and, if engaging in sexual intercourse with a male partner, must agree to use a highly effective method of contraception.
10. Male participants must be surgically sterile for at least 90 days prior to Screening or agree not to donate sperm and, if engaging in sexual intercourse with a female partner who could become pregnant, must agree to use an acceptable method of contraception.

Exclusion Criteria:

1. Clinical signs or symptoms suggestive of polyneuropathy of causes other than CIDP.
2. Known evidence of central demyelination or known history of myelopathy.
3. History or presence of significant medical/surgical condition including any acute illness or major surgery considered to be clinically significant or that could have a potential impact on safety/efficacy or study procedures.
4. Any other condition, including mental illness or prior therapy that would make the participant unsuitable for this study.
5. Known complement deficiency or history of positive titer for anti-C1 antibodies.
6. Diagnosis of systemic lupus erythematosus (SLE) or family history of SLE (defined as a parent, sibling, or child).
7. Participants with an autoimmune disease affecting joints, muscle or nervous system.
8. Any coexisting or overlapping condition, which may interfere with outcome assessments, such as severe diabetic neuropathy, fibromyalgia, inflammatory arthritis or osteoarthritis affecting the hands and feet.
9. Prior history of N. meningitidis infection.
10. History of active malignancy within 5 years prior to screening, except basal cell carcinoma of the skin, curatively resected squamous cell carcinoma of the skin, cervical carcinoma in situ curatively treated or low-grade prostate adenocarcinoma for which appropriate management is observation alone.
11. Positive test results for active human immunodeficiency virus (HIV-1 or HIV-2), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Part B: Time From First Dose to Relapse as Assessed by the Adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) | Part B baseline to Part B end of treatment period (up to Week 52)
  Adjusted INCAT scores range from 0-10 with a score of 10 indicating the greatest degree of disability. A relapse is defined as an increase of ≥1 point from baseline in adjusted INCAT score.

SECONDARY OUTCOMES:
Part B: Time to Decrease of ≥ 4 Points (Centile Metric) in Inflammatory Rasch-built Overall Disability Scale (I-RODS) Score | Part B baseline to Part B end of treatment period (up to Week 52)
  The I-RODS score ranges from 0-100, with lower scores indicating the greatest degree of disability.
Part B: Time to Decrease of ≥ 8 kilopascal (kPa) in Grip Strength in the Dominant Hand | Part B baseline to Part B end of treatment period (up to Week 52)
  This is measured with a handheld device called a vigorimeter.
Part B: Percentage of Participants who Relapse as Assessed by the Adjusted INCAT | Part B baseline to end of treatment period for Part B (up to Week 52)
  Adjusted INCAT scores range from 0-10 with a score of 10 indicating the greatest degree of disability. A relapse is defined as an increase of ≥1 point from baseline in adjusted INCAT score.
Parts A and B: Change in I-RODS Score | Part A baseline up to Part A end of treatment period (up to Week 13); Part A baseline to Part B end of treatment period (up to Part B Week 52)
  The I-RODS score ranges from 0-100, with lower scores indicating the greatest degree of disability.
Parts A and B: Change in Grip Strength in the Dominant Hand | Part A baseline to Part A end of treatment period (up to Week 13); Part A baseline to Part B end of treatment period (up to Part B Week 52)
  This is measured with a handheld device called a vigorimeter.
Parts A and B: Change in Adjusted INCAT Score | Part A baseline to Part A end of treatment period (up to Week 13); Part B baseline to Part B end of treatment period (up to Week 52); Part A baseline to Part B end of treatment period (up to Part B Week 52)
  Adjusted INCAT scores range from 0-10 with a score of 10 indicating the greatest degree of disability.
Parts A and B: Change in Grip Strength in the Nondominant Hand | Part A baseline to Part A end of treatment period (up to Week 13); Part B baseline to Part B end of treatment period (up to Week 52); Part A baseline to Part B end of treatment period (up to Part B Week 52)
  This is measured with a handheld device called a vigorimeter.
Parts A and B: Change in Medical Research Council Sum Score (MRC-SS) | Part A baseline to Part A end of treatment period (up to Week 13); Part B baseline to Part B end of treatment period (up to Week 52); Part A baseline to Part B end of treatment period (up to Part B Week 52)
  The MRC-SS ranges from 0 to 60 with a lower score indicating greater muscle weakness.
Part A: Percentage of Participants with a Confirmed Response to DNTH103 as Assessed by the Adjusted INCAT | Part A baseline to Part A end of treatment period (up to Week 13)
  Adjusted INCAT scores range from 0-10 with a score of 10 indicating the greatest degree of disability. A response is defined as a decrease of ≥1 point from baseline in adjusted INCAT score.
Parts A and B: Change in Euro-Quality of Life Visual Analogue Scale (EQ-VAS) | Part A baseline to Part A end of treatment period (up to Week 13); Part B baseline to Part B end of treatment period (up to Week 52); Part A baseline to Part B end of treatment period (up to Part B Week 52)
  Participants mark their health status from 0 to 100 with 100 indicating the best health state.
Parts A and B: Change in Fatigue Severity Scale (FSS) | Part A baseline to Part A end of treatment period (up to Week 13); Part B baseline to Part B end of treatment period (up to Week 52); Part A baseline to Part B end of treatment period (up to Part B Week 52)
  FSS assesses disabling fatigue in participants with chronic illness.
Parts A and B and OLE: Change in Adjusted INCAT Score | Part A baseline to OLE Week 52 and Week 104; Part B baseline to OLE Week 52 and Week 104; OLE baseline to OLE Week 52 and Week 104
  Adjusted INCAT scores range from 0-10 with a score of 10 indicating the greatest degree of disability.
Part B and OLE: Percentage of Participants With a Confirmed Relapse as Assessed by the Adjusted INCAT | Part B baseline to OLE Week 52 and Week 104; OLE baseline to OLE Week 52 and Week 104
  Adjusted INCAT scores range from 0-10 with a score of 10 indicating the greatest degree of disability. A relapse is defined as an increase of ≥1 point from baseline in adjusted INCAT score.
Parts A, B, OLE, and Safety Follow-up: Number of Participants with Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (SAEs) | Part A baseline through Safety Follow-up period (up to approximately 209 weeks)
  An adverse event (AE) is any undesirable experience associated with the use of a medicine, which does not necessarily have a causal relationship with the medicine. A TEAE is an AE with onset after the start of the medicine, or any worsening of a pre-existing medical condition/AE after the start of the medicine. An SAE is an AE that can cause disability, is life-threatening, results in hospitalization or death, or is a birth defect.
Parts A, B, OLE, and Safety Follow-up: Serum Concentrations of DNTH103 | Part A baseline through Safety Follow-up period (up to approximately 209 weeks)
  Blood samples will be collected for measurement of serum concentrations of DNTH103 at various timepoints both pre- and post-dose.
Parts A, B, and OLE: Change from Baseline in Complement Total Blood Test (CH50) | Part A baseline through Safety Follow-up period (up to approximately 209 weeks)
  Blood samples will be collected to determine changes in CH50 at various timepoints.
Parts A, B, OLE, and Safety Follow-up: Incidence and Titer of Antidrug Antibodies (ADAs) | Part A baseline through Safety Follow-up period (up to approximately 209 weeks)
  Blood samples will be collected to measure ADA against DNTH103 at various timepoints.

CONTACTS AND LOCATIONS:
Locations (114):
- United States (27):
  - Clinical Study Site, Birmingham, Alabama
  - Clinical Study Site, Phoenix, Arizona
  - Clinical Study Site, Scottsdale, Arizona
  - Clinical Study Site, Los Angeles, California
  - Clinical Study Site, San Francisco, California
  - Clinical Study Site, Washington D.C., District of Columbia
  - Clinical Study Site, Maitland, Florida
  - Clinical Study Site, Tampa, Florida
  - Clinical Study Site, Honolulu, Hawaii
  - Clinical Study Site, Chicago, Illinois
  - Clinical Study Site, Edwardsville, Illinois
  - Clinical Study Site, Indianapolis, Indiana
  - Clinical Study Site, Kansas City, Kansas
  - Clinical Study Site, Burlington, Massachusetts
  - Clinical Study Site, East Lansing, Michigan
  - Clinical Study Site, Omaha, Nebraska
  - Clinical Study Site, New York, New York
  - Clinical Study Site, Cincinnati, Ohio
  - Clinical Study Site, Columbus, Ohio
  - Clinical Study Site, Portland, Oregon
  - Clinical Study Site, Dallas, Texas
  - Clinical Study Site, Denton, Texas
  - Cinical Study Site, Houston, Texas
  - Texas Locations, Houston, Texas
  - Clinical Study Site, Round Rock, Texas
  - Clinical Study Site, Sugar Land, Texas
  - Clinical Study Site, Seattle, Washington
- Argentina (7):
  - Cinical Study Site, Buenos Aires, Buenos Aires
  - Cinical Study Site #3, Buenos Aires
  - Cinical Study Site #4, Buenos Aires
  - Clinical Study Site #2, Buenos Aires
  - Clinical Study Site, Buenos Aires
  - Cinical Study Site #2, San Miguel de Tucumán
  - Clinical Study Site, San Miguel de Tucumán
- Australia (2):
  - Clinical Study Site, Randwick, New South Wales
  - Clinical Study Site, Melbourne, Victoria
- Brazil (4):
  - Cinical Study Site, Rio de Janeiro, Rio de Janeiro
  - Cinical Study Site, Natal
  - Cinical Study Site, Salvador
  - Cinical Study Site, São Paulo
- Bulgaria (2):
  - Cinical Study Site, Sofia
  - Clinical Study Site, Sofia
- China (16):
  - Clinical Study Site, Hefei, Anhui
  - Clinical Study Site, Guangzhou, Guangdong
  - Clinical Study Site, Changsha, Hu'Nan
  - Clinical Study Site, Wuhan, Hubei
  - Clinical Study Site, Chifeng, Inner Mongolia
  - Clinical Study Site, Suzhou, Jiangsu
  - Clinical Study Site, Beijing
  - Clinical Study Site, Chengdu
  - Clinical Study Site, Fujian
  - Clinical Study Site, Guangdong
  - Clinical Study Site, Guangzhou
  - Clinical Study Site, Jilin
  - Clinical Study Site, Shanghai
  - Clinical Study Site, Sichuan
  - Clinical Study Site, Taiyuan
  - Clinical Study Site, Wuhan
- Denmark (2):
  - Clinical Study Site, Aarhus
  - Clinical Study Site, Copenhagen
- France (11):
  - Clinical Study Site, Bordeaux
  - Cinical Study Site, Brest
  - Clinical Study Site, Bron
  - Clinical Study Site, Clermont-Ferrand
  - Clinical Study Site, Libourne
  - Clinical Study Site, Marseille
  - Clinical Study Site, Nice
  - Clinical Study Site, Paris
  - Clinical Study Site, Strasbourg
  - Cinical Study Site, Tours
  - Clinical Study Site, Tours
- Clinical Study Site, Tbilisi, Georgia
- Germany (5):
  - Clinical Study Site, Sande, Lower Saxony
  - Clinical Study Site, Aachen
  - Cinical Study Site, Greifswald
  - Clinical Study Site, Rüdersdorf
  - Clinical Study Site, Sande
- Italy (9):
  - Clinical Study Site, Bergamo
  - Clinical Study Site, Bologna
  - Cinical Study Site, Genova
  - Cinical Study Site, Gussago
  - Cinical Study Site, Milan
  - Clinical Study Site, Pavia
  - Clinical Study Site, Ponderano
  - Clinical Study Site, Roma
  - Clinical Study Site #2, Roma
- Latvia (2):
  - Cinical Study Site, Riga
  - Clinical Study Site, Riga
- Malaysia (3):
  - Cinical Study Site, George Town
  - Cinical Study Site, Johor Bahru
  - Cinical Study Site, Kuala Lumpur
- Cinical Study Site, Utrecht, Netherlands
- Poland (5):
  - Clinical Study Site, Bydgoszcz
  - Clinical Study Site, Krakow
  - Clinical Study Site, Lublin
  - Cinical Study Site, Warsaw
  - Clinical Study Site, Wroclaw
- Clinical Study Site, Bucharest, Romania
- Serbia (4):
  - Cinical Study Site, Belgrade
  - Clinical Study Site, Belgrade
  - Clinical Study Site, Kragujevac
  - Clinical Study Site, Niš
- South Korea (6):
  - Cinical Study Site, Daegu
  - Cinical Study Site, Daejeon
  - Cinical Study Site #2, Seoul
  - Cinical Study Site #3, Seoul
  - Cinical Study Site, Seoul
  - Cinical Study Site, Yangsan
- Spain (5):
  - Clinical Study Site, Barcelona, Barcelona
  - Clinical Study Site, Alicante
  - Clinical Study Site, Barcelona
  - Cinical Study Site, Barcelona
  - Clinical Study Site, Bilbao
- Clinical Study Site, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No